CLINICAL TRIAL: NCT06658834
Title: A Multicenter Interventional Study of Romiplostim N01 Combined With Glucocorticoids as the First-line Treatment for Newly Diagnosed Adult Patients With ITP
Brief Title: A Study of Romiplostim N01 as the First-line Treatment for Newly Diagnosed Adult Patients With ITP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other); Weifang People's Hospital (Other); Shenzhen Second People's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Changzhi Medical College (Other); Affiliated Hospital of Nantong University (Other); The First People's Hospital of Yunnan (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Suining Central Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); North China University of Science and Technology (Other); Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024046
Record Dates: First submitted 2024-09-19; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-04

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: ITP; Romiplostim; Continuous Remission
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- romiplostim combined with glucocorticoids (Experimental): Dexamethasone (HD-DXM) at a dose of 40mg/d for 4 days constitutes one cycle. If there is no response on the 10th day, repeat it once. The administration can be either oral or intravenous. Meanwhile, romiplostim N01 is administered with an initial dose of 3µg/kg by subcutaneous injection once a week for up to 6 months.
  Interventions: Drug: Dexamethasone Combined with romiplostim N01
- glucocorticoids (Active Comparator): Dexamethasone (HD-DXM) 40mg/d × 4 days, one cycle. If there is no response on the 10th day, repeat once, administered either orally or intravenously.
  Interventions: Drug: Dexamethasone monotherapy

INTERVENTIONS:
Drug: Dexamethasone Combined with romiplostim N01 — Dexamethasone (HD-DXM) at a dose of 40mg/d for 4 days constitutes one cycle. If there is no response on the 10th day, repeat it once. The administration can be either oral or intravenous. Meanwhile, romiplostim N01 is administered with an initial dose of 3µg/kg by subcutaneous injection once a week for up to 6 months.
  Arms: romiplostim combined with glucocorticoids
Drug: Dexamethasone monotherapy — Dexamethasone (HD-DXM) 40mg/d × 4 days, one cycle. If there is no response on the 10th day, repeat once, administered either orally or intravenously.
  Arms: glucocorticoids

SUMMARY:
This study is a multicenter interventional research on the first-line treatment of newly diagnosed adult patients with immune thrombocytopenia (ITP) using romiplostim N01 in combination with glucocorticoids. The primary endpoint of this study is to assess the efficacy of romiplostim N01 combined with glucocorticoids in untreated newly diagnosed adult ITP patients after 6 months of administration.

The subjects will be divided into the experimental group and the control group for treatment.

Experimental group: Dexamethasone (HD-DXM) 40mg/d × 4 days, one cycle. If there is no response on the 10th day, repeat once, administered either orally or intravenously. Simultaneously, romiplostim N01 is administered at an initial dose of 3µg/kg, by subcutaneous injection, once a week, for a maximum of 6 months.

Control group: Dexamethasone (HD-DXM) 40mg/d × 4 days, one cycle. If there is no response on the 10th day, repeat once, administered either orally or intravenously.

DETAILED DESCRIPTION:
This study is a multicenter interventional research, and it is planned to incorporate 129 newly diagnosed adult ITP patients who have not undergone treatment.

For patients meeting the inclusion criteria, after signing the informed consent and passing the screening, they will be randomly grouped.

The study encompasses a screening period (from the signing of the informed consent form by the subject to before the first administration of the drug), a treatment period (including dexamethasone monotherapy and combined treatment of dexamethasone and romiplostim N01), and a follow-up period.

Screening period: Assess the inclusion and exclusion criteria. Those who fulfill the conditions can enter the treatment period.

Treatment period: Baseline visits are conducted for the screened eligible subjects, and they are randomly assigned to the experimental group and the control group at a ratio of 2:1.

Administration protocol:

Experimental group: Dexamethasone (HD-DXM) 40mg/d × 4d, one cycle. If there is no response on the 10th day, repeat once, administered orally or intravenously. Simultaneously, romiplostim N01 is administered, with an initial dose of 3µg/kg, by subcutaneous injection once a week, for up to 6 months.

Control group: Dexamethasone (HD-DXM) 40mg/d × 4d, one cycle. If there is no response on the 10th day, repeat once, administered orally or intravenously.

*Dosage of romiplostim N01: The initial dose is 3µg/kg and can be initiated within 4 days of dexamethasone treatment.

When the platelet count is < 50 × 10^9/L, the patient will receive an increment in the dose of romiplostim N01 by 2µg/kg weekly, with a maximum dose of 10µg/kg. When 200 × 10^9/L > platelet count ≥ 50 × 10^9/L, the administration dosage remains unchanged. When 400 × 10^9/L > platelet count ≥ 200 × 10^9/L for two consecutive weeks, the dose is reduced by 1µg/kg. When the platelet count is ≥ 400 × 10^9/L, discontinue the drug. When the platelet count < 200 × 10^9/L, resume administration, and the administration dose is 1µg/kg less than before drug cessation.

Follow-up period: Enter the follow-up period after the conclusion of treatment. Follow-up: Collect all adverse events (AEs) considered related to the study drug, follow up until the 14th week after the end of treatment, through clinical follow-up or telephone follow-up, and collect information on AEs, concomitant medications and concomitant treatments of the subjects. The researcher can increase the number of visits as necessary for AE follow-up to monitor the alleviation of AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the written informed consent form before enrollment;
2. Age ranging from 18 to 75 years old;
3. Be clinically diagnosed with primary immune thrombocytopenia for less than 3 months before randomization;
4. Have not received splenectomy or at least one first-line ITP treatment or emergency treatment in the past;
5. Have not received romiplostim treatment;
6. ECOG PS score: 0 - 2;
7. Platelet value < 30×10^9/L;
8. The expected survival period at the screening is ≥ 12 weeks;
9. For subjects of reproductive age, agree to take reliable contraceptive measures throughout the study period (including male or female condoms, contraceptive foams, contraceptive gels, contraceptive membranes, contraceptive ointments, contraceptive suppositories, abstinence, and intrauterine device placement, etc.); Female subjects who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation or menopause for more than 1 year, and male subjects who have undergone bilateral vasectomy or ligation are excluded;
10. Voluntarily join this study, sign the informed consent form, and have good compliance.

Exclusion Criteria:

1. Suffering from other hematopoietic system diseases except ITP, including but not limited to leukemia, thrombocytopenia caused by tumor treatment, myeloproliferative diseases, multiple myeloma and myelodysplastic syndrome, etc.;
2. Having undergone splenectomy before the first administration;
3. Having received ITP drug treatment (including emergency treatment) before the first administration;
4. Having used drugs with c-Mpl (thrombopoietin receptor) stimulating effects within 4 weeks before the first administration;
5. Having received hematopoietic growth factor preparations (such as granulocyte colony-stimulating factor, macrophage colony-stimulating factor, erythropoietin, interleukin-11, etc.) within 4 weeks before the first administration;
6. Having received antibody drugs (such as rituximab, etc.) within 14 weeks before the first administration;
7. Having received any Chinese herbal medicine or nutritional supplement (except vitamin supplements and mineral supplements) for the purpose of increasing platelets within 1 week before the first administration;
8. Having been diagnosed with arterial thrombosis (such as cerebral thrombosis, transient ischemic attack or myocardial infarction), or having a history or complication of venous thrombosis (such as deep vein thrombosis, pulmonary embolism), or using anticoagulants or antiplatelet drugs at the beginning of screening;
9. Having a history of severe cardiovascular diseases (such as grade III/IV congestive heart failure, arrhythmia or angina pectoris that increases the risk of thromboembolic events, unstable angina pectoris, having undergone coronary artery stent implantation, angioplasty or coronary artery bypass grafting);
10. Secondary thrombocytopenia caused by autoimmune diseases such as antiphospholipid antibody syndrome, systemic lupus erythematosus, Hashimoto's thyroiditis, Even's syndrome and Sjogren's syndrome;
11. Positive results for either human immunodeficiency virus antibody or syphilis antibody screening; positive hepatitis C antibody and HCV-RNA exceeding the upper limit of the study center's laboratory test; positive hepatitis B surface antigen and HBV-DNA exceeding the upper limit of the study center's laboratory test;
12. Having participated in other clinical studies within 3 months before the first administration;
13. Being pregnant or lactating, or having a pregnancy plan;
14. Having fertility and being judged by the researcher as not fully adopting contraceptive measures;
15. Having a history of severe drug allergic reactions or being known to be allergic to glucocorticoids or Nplate® (romiplostim) or the components of QL0911;
16. Unable to comply for mental reasons;
17. Judged by the researcher as not suitable to participate in this trial;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with continuous remission. | 6 months
  Continuous remission is defined as the maintenance of the therapeutic effect of patients for at least 6 months since achieving remission, without the need for additional ITP-specific treatment.

SECONDARY OUTCOMES:
The total effective rate GR | 6 months
  The total effective rate GR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Effective R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms).
The proportion of patients with the initial response (reaching the effective standard within one month of the start of treatment) | one month of the start of treatment
  The total effective rate GR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Effective R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms within one month).
The proportion of patients reaching the effective standard 3 months after the start of treatment. | 3 months after the start of treatment
  The total effective rate GR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Effective R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms within 3 month).
The proportion of patients reaching the effective standard 6 months after the start | 6 months after the start
  The total effective rate GR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Effective R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms within 6 month).
The maximum consecutive weeks of platelet response | 6 months
  The consecutive weeks with platelet count > 30×10^9/L in the absence of any rescue treatment. Adverse events (evaluated using Version 5.0 of the "Common Terminology Criteria for Adverse Events (NCI CTC AE)") etc.
The proportion of subjects receiving rescue treatment. | 6 months
  The proportion of subjects receiving rescue treatment.
According to the WHO bleeding score standard, the incidence and severity of bleeding symptoms. | 6 months
  According to the WHO bleeding score standard, the incidence and severity of bleeding symptoms.
Adverse events | 6 months
  evaluated using Version 5.0 of the "Common Terminology Criteria for Adverse Events (NCI CTC AE)".

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China